CLINICAL TRIAL: NCT01035398
Title: Molecular Epidemiology of Esophageal Cancer: Pilot Project
Brief Title: Genetic and Environmental Risk Factors Related to Esophageal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Christopher Christiani, Pulmonary Associate, Massachusetts General Hospital
Other Study IDs: CDR0000450143; MGH-1999-P-010178/23 (Other: Partners IRB); 5R01CA109193-04 (NIH)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Cancer
Keywords: stage 0 esophageal cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Gathering information about genes, cigarette smoking, and diet may help doctors learn more about risk factors that may cause esophageal cancer.

PURPOSE: This clinical trial is studying genetic and environmental risk factors related to esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the role of several genetically-determined factors in combination with cigarette smoking and diet in the etiology and prevention of esophageal cancer.
* Identify polymorphisms in metabolizing enzymes (e.g., phase I or II metabolism [GSTM1, GSTT1,CYP1A1, CYP3A5, mEH, NQO1, GSTP1], DNA repair [XRCC1, ERCC2], free-radical formation [MPO, MnSOD], inflammatory genes [ IL1-beta], metastatic potential [MMP1], and cell cycle or tumor suppression [p21, p53]) and related path genes of susceptibility for esophageal cancer.

OUTLINE: Blood and tumor tissue samples are collected. DNA purified from these samples is analyzed using DNA-based assays to determine polymorphisms in various related gene pathways.

Patients complete questionnaires concerning environmental, smoking and diet habits.

PROJECTED ACCRUAL: A total of 1,000 tissue samples from patients and healthy participants (750 patients and 250 healthy participants) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of esophageal cancer (patient)

    * Newly diagnosed disease
    * Receiving care at Massachusetts General Hospital, Thoracic Oncology Center
  * Friend or spouse of patient (healthy participants)

PATIENT CHARACTERISTICS:

* No concurrent psychiatric incapacity or dementia

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2000-04; Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Polymorphisms in various pathways, DNA repair, free-radical formation, inflammatory genes, metastatic potential, and cell cycle or tumor suppression in blood samples | 2000-2016
Comparison of presence or absence of variant polymorphisms between cases and controls | 2000-2016
Correlation between polymorphisms in blood samples and polymorphisms in tissue specimens | 2000-2016
Analyses of dietary factors and Helicobacter pylori infection (previous vs current) | 2000-2016

CONTACTS AND LOCATIONS:
Overall Officials: David C. Christiani, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard School of Public Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No